CLINICAL TRIAL: NCT03537183
Title: Will Elevated Left Ventricle Filling Pressures Decrease by a Group Exercise Program in Patients With Hypertrophic CardioMyopathy? - A Randomized Clinical Trial
Brief Title: Will Elevated Left Ventricle Filling Pressures Decrease by a Group Exercise Program in Patients With Hypertrophic CardioMyopathy?
Acronym: WEDGE-HCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Helga Gudmundsdottir, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 63446
Record Dates: First submitted 2018-05-09; First posted 2018-05-25 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: hypertrophic cardiomyopathy; exercise training; PCWP
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual activity level (No Intervention): 12 weeks of usual activity level
- Exercise training (Active Comparator): 12 weeks of moderate intensity exercise training, 3 hours a week
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — 12 weeks, 3 hours a week, moderate intensity exercise training
  Arms: Exercise training

SUMMARY:
Aims and objectives: The primary objective of this study is to assess whether a structured exercise program improves cardiac relaxing properties in patients with hypertrophic cardiomyopathy (HCM).

Background: HCM is a hereditary disease in which the myocardium becomes thickened without an identifiable cause (other than genetic). It is the most common genetic cardiovascular disease with an estimated prevalence of 1/500 (i.e. 10.000 affected individuals in Denmark). The majority of patients with HCM suffers from shortness of breath and reduced exercise capacity due to increased left ventricular (LV) stiffness. Exercise training has been shown to improve exercise capacity and symptoms in patients with HCM, but the mechanisms responsible for this improvement are not known.

Methods and materials: The study is a randomized, single blinded, prospective, controlled clinical trial. Eighty patients are recruited from outpatient clinics in the Capital Region of Denmark. Patients are randomized in a 1:1 ratio to 12 week of moderate-intensity exercise training or usual activity level. Assessments will include right heart catheterization, echocardiography, cardiopulmonary exercise testing, blood-samples, quality of life, and, in a subgroup of patients, cardiac magnetic resonance imaging. The primary end-point is change in LV filling pressure assessed as pulmonary capillary wedge pressure at 25 W workload.

Expected outcome and perspectives: The investigators hypothesize that an exercise training program will reduce cardiac stiffness and improve symptoms in patients with HCM. Training of HCM patients has long been debated and the topic is poorly researched. The effects of exercise on hemodynamics in HCM patients are unknown and a better understanding of these mechanisms is pivotal for improving treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years at the time of screening
2. Documented phenotypic HCM (maximal wall thickness ≥15mm, or ≥13mm in a first degree relative with a definite or likely disease causing genetic mutation (appendix 1)
3. Not exercising regularly (dedicated moderate or high-intensity exercise >1 hour weekly)
4. NYHA class I-IV.

Exclusion Criteria:

1. Phenocopies (i.e. syndromes, metabolic disorders (appendix 2))
2. A history of exercise induced syncope within the last year, severe angina (CCS III-IV), hemodynamically severe valvular disorders
3. Scheduled septal reduction therapy, less than 3 months after septal reduction therapy or known LVOT gradient above 30 mmHg at rest
4. Severe hypertension (Systolic blood pressure >200 mmHg or diastolic blood pressure >110 mmHg).
5. Inability to exercise due to orthopedic or other non-cardiovascular limitations.
6. Pregnancy
7. Changes in medication that may affect exercise capacity and/or hemodynamics (i.e. beta blockers and calcium channel blockers)
8. Any condition (eg, psychiatric illness) or situation that, in the investigator's opinion, could put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to follow-up in PCWP at 25 W | 12 weeks
  Pulmonary capillary wedge pressure (mmHg)

SECONDARY OUTCOMES:
Pulmonary capillary wedge pressure | 12 weeks
  At rest, at 25% and 50% of the maximum workload and at maximum workload ( measured as mmHg)
Workload adjusted Pulmonary capillary wedge pressure | 12 weeks
  At rest, at 25% and 50% of the maximum workload and at maximum workload, measured as mmHg/kg/W
Systemic vascular resistance | 12 weeks
  Resting and exercise systemic vascular resistance at rest, 25 W, 25% and 50% of the maximum workload and at maximum workload ( measured as mmHg)
Exercise capacity | 12 weeks
  Measured as watt at maximum workload
Heart rate | 12 weeks
  At rest, during exercise and at maximum exercise capacity (beats/min)
Blood pressure | 12 weeks
  At rest, at maximum workload, 6 minutes after cease of workload (mmHg)
Cardiac index | 12 weeks
  At rest, 25W and at maximum workload (L/min/m2):
Arterio-venous difference | 12 weeks
  At rest, 25W and at maximum workload (ml O2/L)and workload corrected (mlO2/L/W)
VO2 max | 12 weeks
  Measered as ml O2/min/kg
Quality of life questionnaire | 12 weeks
  Measured by Kansas City Cardiomyopathy score
NT-Pro-BNP | 12 weeks
  (pmol/L)
Troponin-T | 12 weeks
  (mmol/L)
Echocardiographic parameters | 12 weeks
  At rest: E/e'-ratio, E/A-ratio, deceleration time, LVOT gradient (mmHg). During exercise from 25W to maximum workload: E/e'-ratio, E/A-ratio, deceleration time, LVOT gradient(mmHg).

OTHER OUTCOMES:
Left ventricular fibrosis | 12 weeks
  (assessed as late gadolinum enhancement) and extracellular volume (assessed using T1-mapping) will be assessed in the subgroup of patients without contraindications to CMR and will be correlated to LV filling pressures.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Gudmundsdottir HL, Axelsson Raja A, Rossing K, Rasmusen H, Snoer M, Andersen LJ, Gottlieb R, Christensen AH, Bundgaard H, Gustafsson F, Thune JJ. Exercise Training in Patients With Hypertrophic Cardiomyopathy Without Left Ventricular Outflow Tract Obstruction: A Randomized Clinical Trial. Circulation. 2025 Jan 14;151(2):132-144. doi: 10.1161/CIRCULATIONAHA.124.070064. Epub 2024 Nov 8. PMID 39513255